CLINICAL TRIAL: NCT05560347
Title: The Effect of Hot Water Application on Pain, Comfort and Vital Singns After Cesarean
Brief Title: The Effect of Hot Water After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tugba Sivri, Graduate Student, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0920211278
Record Dates: First submitted 2022-09-20; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Cesarean Section
Keywords: Cesarean section; Hot Water; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, experimental, clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Hot water will be applied to the participants in the experimental group at the 2nd and 6th hours postoperatively. During the hot water application, the feet of the individual will be immersed in the hot water application device and kept in the device for 20 minutes. At the end of the 20th minute, the feet of the individual will be removed from the device and dried with a towel for 10 minutes and the application will be completed. The data will be obtained by using the Introductory Information Form, Visual Analog Scale (VAS), Postpartum Comfort Scale and Post Cesarean Patient Evaluation Form.
  Interventions: Other: Hot water application
- Control Group (No Intervention): Routine care will be given to the control group

INTERVENTIONS:
Other: Hot water application — Hot application is applied by contacting any part of the body with a temperature of 40-45 degrees. Hot application stimulates the touch receptors and has a vasodilation effect. Thermoreceptors in the foot are stimulated by applying heat to the feet, and this stimulation is thought to be effective in reducing the activation of the sympathetic nervous system and thus reducing pain.
  Arms: Experimental Group

SUMMARY:
The main subject of this project is the problem of pain after cesarean section. It is known that the application of hot water reduces the pain of the patients, with the decrease of the pain, the vital signs of the patient are improved and the comfort level increases. Our project work is based on this subject.

DETAILED DESCRIPTION:
Cesarean section surgery is an attempt to become mandatory and applied in cases where vaginal delivery is dangerous for the mother and fetus. One of the most common problems that women experience in the process after cesarean section is pain. This pain experienced for various reasons such as incision site pain, headache and pain caused by uterine contractions negatively affects the comfort of the woman in the postpartum period. In addition to pain, especially after cesarean section, the woman cannot be mobilized, the presence of a urinary catheter, the negative effects caused by anesthesia cause the mother to be unable to meet her own self-care needs and perform life activities, which disrupts the comfort of the woman As a result of the study in which Çankaya evaluated the comfort of mothers who gave birth by cesarean section, it was found that 78% of mothers have pain at the incision site and this negatively affects maternal comfort The pain that cannot be controlled causes a limitation in activities, respiratory, circulatory and digestive system problems in the postoperative period and prolongs the recovery period. Therefore, the woman's pain should be managed and aimed at minimizing it. In this context, when looking at the literature, it is noticeable that there are various methods of dealing with pain after cesarean section. Pharmacological treatment options are preferred in the management of pain after cesarean section due to their ability to reduce and treat pain in a shorter period of time. After cesarean section, more often non-steroidal anti-inflammatory drugs or paracetamol-derived drugs are used. Non-pharmacological methods should also be used in pain management to support pharmacological methods and minimize the use of analgesics Some non-pharmacological methods used can be listed as follows; aromatherapy, massage hand/foot massage, listening to music, progressive relaxation exercises, acupuncture, hot and cold applications. A limited number of studies on hot application have been found in the literature. Based on these results, this study is planned to examine the effects of hot water application on pain comfort and life signs.

ELIGIBILITY:
Inclusion Criteria

* At least primary school graduate
* 18 years and older
* No history of chronic disease (Diabetes, etc.)
* Risky pregnancy (Premature rupture of membranes, Premature birth threat, preeclampsia etc.) without diagnosis
* Women who do not develop any complications (Atony, abnormal bleeding, need for blood transfusion, risks related to anesthesia, bladder injury, etc.) during or after the operation.

Exclusion Criteria:

* Not a primary school graduate
* Under 18 years old
* Blood pressure, diabetes, etc. sick
* Diagnosed with risky pregnancy,
* Complications developing during or after surgery
* Women who do not want to participate in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in Pain assessed by VAS score | 3rd and 6th hours after cesarean section
  Chancing in pain after cesarean section. The data will be obtained by using Visual Analog Scale. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain.

SECONDARY OUTCOMES:
Change the comfort score | 12 th hours after cesarean section
  Chancing the comfort score after cesarean section. The data will be obtained by using the Postpartum Comfort Scale. Postpartum Comfort Scale (PCS): It is a Likert-type scale consisting of 34 items to determine the postpartum comfort. The lowest and the highest scores in the scale are 34 and 170. It has three sub dimensions; physical, psycho spiritual and sociocultural. Scores close to 170 indicate ahigh level of comfort.

IPD SHARING:
Plan to Share IPD: No